CLINICAL TRIAL: NCT05748639
Title: Randomized Controlled Trial of an Integrated Digital Cognitive-Behavioral Therapy (CBT) and Pharmacotherapy Intervention for Adults With Alcohol Use Disorders
Brief Title: Integrated Digital Intervention for Alcohol Use Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Quit Genius (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QG01
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Practice Management, Medical

STUDY DESIGN:
Intervention Model Description: The study is designed as a 2-arm, parallel-group, randomized controlled trial with 12-, 24-, 36-, and 52-week follow-up, to evaluate the effect of the treatment group (QG-A) versus a control group (MM) on alcohol use outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quit Genius - Alcohol (Experimental): QG-A is a smart phone application targeting alcohol use disorder. QG-A includes standardized cognitive-behavioral therapy in the form of videos, in-app text, audio recordings, and quizzes. The application provides users with information on how to reduce or abstain from alcohol use. Once successfully enrolled in QG-A, a medical provider will evaluate each QG-A participant for appropriateness for pharmacotherapy during an initial 60-minute assessment to confirm an alcohol use disorder diagnosis and collect relevant medical and psychiatric history of the patient. The medical provider will subsequently prescribe oral naltrexone via the QG-A telemedicine platform. A study counselor will provide manualized CBT-based support to QG-A participants via the video telemedicine function, as well as asynchronously via the in-app chat function.
  Interventions: Other: Mobile health application
- Medical Management (Active Comparator): Medical management comprises standard care for alcohol use disorder. A medical provider, upon evaluation of each participant for appropriateness for pharmacotherapy, will subsequently prescribe naltrexone via a non-QG-A telemedicine platform, according to standard clinical practice. Participants will meet with the medical provider monthly over the 6-month course of treatment. In MM, participants receive dose adjustments and brief medical management as normally provided to patients in office-based settings (session duration is 15-20 minutes). The medical provider will deliver education about the study medication and answer any participant questions. Subsequent 15-20 minute sessions will review drinking patterns, overall functioning, medication adherence, and adverse effects. Participants who discontinue medication because of intolerance can continue to attend monthly medical management sessions to support abstinence.
  Interventions: Other: Medical Management

INTERVENTIONS:
Other: Mobile health application — Participants randomized to receive the QG-A (Experimental) intervention will receive monthly appointments with a medical provider, access to naltrexone, and weekly and bi-weekly appointments with a licensed clinical counselor through an integrated digital health application.
  Other Names: QG-A
  Arms: Quit Genius - Alcohol
Other: Medical Management — Participants randomized to receive the MM (Control) intervention will receive monthly appointments with a medical provider and access to naltrexone.
  Other Names: TAU
  Arms: Medical Management

SUMMARY:
This study is a two-arm randomized clinical trial comparing the Quit Genius intervention for alcohol use disorder (QG-A) to usual care (TAU), comprising medical management of alcohol use disorders with pharmacotherapy. Participants (N=300) will be randomly assigned to either QG-A or TAU, and will be assessed at baseline, monthly throughout the 6-month intervention phase and at 3 and 6 months post-treatment, to investigate the impact of QG-A, relative to TAU on alcohol use, psychological symptoms, and health service utilization. The primary aim of the study is to evaluate the efficacy of QG-A, relative to TAU in reducing alcohol use and associated mental health and functional outcomes. A secondary aim is to examine the cost-effectiveness of QG-A, including cost savings and impact on productivity.

DETAILED DESCRIPTION:
Effective and evidence-based therapies are available for management of Alcohol Use Disorder (AUD) with a variety of pharmacological and psychosocial interventions supported by a sizable clinical trials literature. However, a major barrier in addressing this significant public health issue is the fact that a majority of individuals with AUD are not receiving treatment. Evidence shows that Individuals with problematic alcohol use may be dissuaded from seeking help due to a lack of accessibility of services, stigmatization, low motivation, or cost of treatment.

Traditional methods of treating AUD typically utilize a behavioral, pharmacological or a combination approach. Medication-assisted treatment (MAT) is the use of medications, in combination with psychosocial therapies, to provide an integrated approach to the treatment of substance use disorders. The MAT approach to treating AUD has been widely successful, with various combinations of pharmacotherapy and psychosocial interventions showing efficacy in the reduction of alcohol use. In particular, the combination of psychosocial therapies such as CBT, MET and 12 steps have proven highly successful when used in combination with the opioid receptor antagonist Naltrexone (NTX). Yet, a lack of accessibility, practicality and adherence to traditional methods has left many alcohol users without the means to effectively deal with their addictions.

Digital therapeutics can address these issues and provide advantages including anonymity, convenience, accessibility, cost-effectiveness, and privacy. Digital therapies can also target individuals with problematic alcohol use who are in different psychological stages of change, allowing potential users to investigate treatment options without the stigma associated with face-to-face interactions. Additionally, these digitized evidence-based therapies have the potential to increase treatment adherence, and because the content is standardized, it can be delivered with greater consistency than face-to-face therapy, lending itself to a clinical research approach.

Quit Genius Alcohol (QG-A) is a newly developed comprehensive treatment program for AUD, utilizing a combination of a mobile-app, pharmacotherapy, and breath sensor. The mobile app is informed by the principles of CBT, Motivational Enhancement Therapy (MET), and community reinforcement. QG delivers personalized, behavioral support adjunct to proven pharmacotherapies to individuals who are seeking to reduce their alcohol consumption. An initial pilot investigation of QG-A demonstrated the feasibility of the intervention as well as some promising preliminary outcomes with regards to alcohol use and related psychological variables that are recognized mechanisms of change in CBT treatment for addicted populations.

As such, the objective of the proposed investigation is to build on the preliminary outcomes and evaluate the effectiveness of QG-A. This study will compare the efficacy of QG-A, which combines CBT based counseling with pharmacotherapy for alcohol use disorders (naltrexone), delivered via an mobile health app (QG-A), relative to usual care for adults with AUD, which comprises medical management with naltrexone (MM), in reducing alcohol use and associated psychological and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older;
* A US resident;
* Using Apple iPhone (5th generation or higher) or Android phone (version 18 or higher);
* Diagnostic and Statistical Manual-V diagnosis of either a moderate or severe Alcohol Use Disorder;
* Currently has health insurance;
* Able to provide informed consent;
* Currently employed;
* Willing and able to participate in study procedures;
* Willing to take naltrexone; and
* Good general health or, in the case of a medical/psychiatric condition needing ongoing treatment, potential participants should be under the care of a physician or other qualified healthcare provider with whom the participant provides documented permission to coordinate care with the QG-A care team.

Exclusion Criteria:

* Known sensitivity to naltrexone;
* Pregnant, breast feeding, or unwilling to use contraceptive methods;
* Presence of serious medical or psychiatric disorders that would, in the opinion of the medical provider, make participation hazardous or regular follow-up unlikely (e.g., suicidal ideation, acute hepatitis, unstable cardiovascular, liver or renal disease);
* A current pattern of alcohol or sedative use, as assessed by the QG-A licensed medical provider, which would preclude safe participation in the study and/or would likely require imminent medical detoxification;
* Having used acamprosate, disulfiram, or naltrexone, within the past 30 days prior to screening;
* Takes an opioid medication on a routine basis for a pain condition or has anticipated/planned surgery that will require opioid maintenance during the study timeframe;
* Has undergone more than one inpatient medical detoxification treatment; and
* Lack of proficiency in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Alcohol use | Baseline to 6-months post-treatment entry
  Change in past 30-day alcohol use

CONTACTS AND LOCATIONS:
Locations (1):
- Quit Genius, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Result] Bandawar M, Narasimha VL, Chand P. Use of digital technology in addiction disorders. Indian J Psychiatry. 2018 Feb;60(Suppl 4):S534-S540. doi: 10.4103/psychiatry.IndianJPsychiatry_21_18. PMID 29540927
- [Result] Singh K, Drouin K, Newmark LP, Lee J, Faxvaag A, Rozenblum R, Pabo EA, Landman A, Klinger E, Bates DW. Many Mobile Health Apps Target High-Need, High-Cost Populations, But Gaps Remain. Health Aff (Millwood). 2016 Dec 1;35(12):2310-2318. doi: 10.1377/hlthaff.2016.0578. PMID 27920321
- [Result] Messner E-M, Probst T, O'Rourke T, Stoyanov S, Baumeister H. mHealth Applications: Potentials, Limitations, Current Quality and Future Directions. In: Baumeister H, Montag C, eds. Digital Phenotyping and Mobile Sensing: New Developments in Psychoinformatics. Studies in Neuroscience, Psychology and Behavioral Economics. Springer International Publishing; 2019:235-248. doi:10.1007/978-3-030-31620-4_15
- [Result] Kranzler HR, Stephenson JJ, Montejano L, Wang S, Gastfriend DR. Persistence with oral naltrexone for alcohol treatment: implications for health-care utilization. Addiction. 2008 Nov;103(11):1801-8. doi: 10.1111/j.1360-0443.2008.02345.x. PMID 19032530
- [Result] Hammarlund R, Crapanzano KA, Luce L, Mulligan L, Ward KM. Review of the effects of self-stigma and perceived social stigma on the treatment-seeking decisions of individuals with drug- and alcohol-use disorders. Subst Abuse Rehabil. 2018 Nov 23;9:115-136. doi: 10.2147/SAR.S183256. eCollection 2018. PMID 30538599
- [Result] Srisurapanont M, Jarusuraisin N. Naltrexone for the treatment of alcoholism: a meta-analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2005 Jun;8(2):267-80. doi: 10.1017/S1461145704004997. PMID 15850502
- [Result] Miller PM, Book SW, Stewart SH. Medical treatment of alcohol dependence: a systematic review. Int J Psychiatry Med. 2011;42(3):227-66. doi: 10.2190/PM.42.3.b. PMID 22439295